CLINICAL TRIAL: NCT03931304
Title: Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy in Peritoneal Carcinomatosis From Ovarian Cancer
Brief Title: Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy in Peritoneal Carcinomatosis From Ovarian Cancer (Cyto-chip 2)
Acronym: Cyto-chip 2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Cyto-chip 2
Record Dates: First submitted 2018-10-10; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2018-10

CONDITIONS: Peritoneal Carcinoma; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases group: Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure
  Interventions: Procedure: Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure
- Control group: Cytoreductive surgery alone

INTERVENTIONS:
Procedure: Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure — Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure
  Other Names: Cytoreductive surgery alone
  Groups: Cases group

SUMMARY:
Epithelial ovarian carcinoma (EOC) is one of the main cause of death from cancer in women in the Western world. It is often diagnosed at an advanced stage and the disease remains confined to the peritoneal cavity for much of its natural history. Despite a high rate of response to first-line therapy, about 20% of EOC are naturally resistant to platinum and about 2/3 of patients with initial response will recur within 5 years. Most tumour recurrences will develop resistance to systemic platinum over time. The prognosis of these patients with persistent or recurrence disease remains poor despite salvage therapy including alternative systemic chemotherapy and further cytoreductive surgery (CRS). Since twenty years, centers have pursued comprehensive CRS combined with Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for the management of peritoneal surface malignancies (PSM). This combined approach is the standard of care for the management of some rare peritoneal disease such as pseudomyxoma peritonei or peritoneal mesothelioma. EOC should be an ideal target for this loco-regional treatment, as most of its evolution remains confined to intraperitoneal cavity and because of its sensitivity to chemotherapy. Intraperitoneal chemotherapy has been shown to have significant efficacy in frontline EOC in 3 large randomized studies. Recently, French clinical guidelines have been edited to recommend CRS+HIPEC in patients with ovarian, tubal or primitive carcinomatosis FIGOI IIIC, initially not resectable (Grade B). HIPEC adds some advantages to this intraperitoneal chemotherapy: the hyperthermia effect with its direct cytotoxicity demonstrated in vitro, the synergistic effect with some anticancer agents and, the deliverance immediately following CRS, avoiding the problem of "cancer cell entrapment" by postoperative or posttherapeutic adhesions that limits distribution of chemotherapy agents to all sites. The use of HIPEC for EOC was reported into relatively small case-series from single institutions. Results from a single centre cannot be extrapolated to other centres because of the heterogeneity of patient's selection and HIPEC techniques.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed peritoneal carcinomatosis from ovarian cancer
* Metachronous/synchronous peritoneal carcinomatosis
* Grade FIGO (International Federation of Gynecology and Obstetrics) III or IV
* Peritoneal Cancer Index (PCI) available
* Indication for cytoreductive surgery +/- HIPEC
* Complete macroscopic cytoreduction: CCR (cytoreduction score) -0/1

Exclusion Criteria:

* Non complete macroscopic cytoreduction: CCR (cytoreduction score) -2
* Peritoneal mesothelioma, pseudomyxoma peritonei
* Extra peritoneal metastases

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian peritoneal metastases.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of 3-years disease free survival | 3 years
  From the date of cytoreductive surgery with Hyperthermic Intraperitoneal Chemotherapy to death or to the end of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No